CLINICAL TRIAL: NCT07169682
Title: Effects of IL17/23 Inhibitors on Markers of Subclinical Atherosclerosis in Patients With Psoriasis: an Observational Study
Brief Title: Effects of IL17/23 Inhibitors on Markers of Subclinical Atherosclerosis in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Andreas Syggros Hospital of Venereal and Dermatological Diseases (Other)
Responsible Party: Principal Investigator, Aikaterini Tsiogka, dermatologist, clinical research associate, National and Kapodistrian University of Athens
Other Study IDs: 3610/20-05-2021
Record Dates: First submitted 2025-08-27; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis; Cardiovascular Disease; Atherosclerosis
Keywords: psoriasis; atherosclerosis; cardiovascular disease; psoriatic arthritis
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases; Atherosclerosis; Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: IL17 inhibitor
  Interventions: Drug: interleukin 17 inhibitor
- Group 2: IL23 inhibitor
  Interventions: Drug: interleukin-23 inhibitor
- Group 3: conventional systemic agent or apremilast
  Interventions: Drug: conventional systemic agent or apremilast

INTERVENTIONS:
Drug: interleukin 17 inhibitor — 52 weeks
  Groups: Group 1
Drug: interleukin-23 inhibitor — 52 weeks
  Groups: Group 2
Drug: conventional systemic agent or apremilast — 52 weeks
  Groups: Group 3

SUMMARY:
Data on the antiatherogenic effect of IL23 inhibitors are sparse. This study aimed to assess the impact of one-year treatment with an IL17 or IL23 inhibitor on arterial stiffness in patients with moderate-to-severe psoriasis.

This observational cohort study included patients with moderate-to-severe psoriasis treated with either an IL17 inhibitor or an IL23 inhibitor or a conventional systemic agent/apremilast (control group) for 52 weeks. The primary outcome was the evaluation of changes in carotid-femoral pulse wave velocity (PWV) and augmentation index normalized to 75 beats/min (AIx75) after 24 and 52 weeks. Secondary outcomes were the comparison of change in PWV and AIx75 between the study groups and the assessment of psoriasis disease severity scores and in ankle-brachial index (ABI).

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe psoriasis (Psoriasis Area Severity Index (PASI) score > 10 or Body Surface Area (BSA) >10 or Dermatology Life Quality Index (DLQI) >10)
* Indication for treatment with an IL17 or an IL23 inhibitor based on disease characteristics and comorbidities

Exclusion Criteria:

* Prior treatment with an IL17 or an IL23 inhibitor
* Prior therapy with an TNFa-inhibitor for up to 3 months before entering the study
* Chronic or severe acute infections, malignancy
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with plaque psoriasis with or without psoriatic arthritis, who were monitored in the outpatient department for psoriasis of "Andreas Syngros" hospital for skin diseases and were planed to start treatment with an IL17 inhibitor or an IL23 inhibitor on a conventional systemic agent/apremilast
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
change of pulse wave velocity (PWV) from baseline to week 24 and 52 | from enrollment to the end of treatment at week 52
  PWV can range from approximately 6.6 m/s in patients under 30 to 11.7 m/s in patients over 70 years of age; higher scores mean a worse outcome
change of augmentation index normalized to 75 beats/min (AIx75) from baseline to week 24 and 52 | from enrollment to the end of treatment at week 52
  no single universally accepted normal range for an AIx@75; lower values indicate better arterial health, with values below 20-25% often considered optimal, and values above 30% associated with increased arterial stiffness and cardiovascular risk

SECONDARY OUTCOMES:
comparison of change in PWV between the study groups | From enrollment to the end of treatment at 52 weeks
change in psoriasis area severity index (PASI) | From enrollment to the end of treatment at 52 weeks
  range 0-72; higher scores mean a worse outcome
change in ankle-brachial index (ABI) | From enrollment to the end of treatment at 52 weeks
  range 0.9-1.4; higher scores mean worse outcome
comparison of change in AIx75 between the study groups | from enrollment to the end of treatment at 52 weeks
change in body surface area (BSA) | From enrollment to the end of treatment at 52 weeks
  values 0-100%, higher scores mean a worse outcome
change in physician's global assessment (PGA) | From enrollment to the end of treatment at 52 weeks
  range 0-5; higher scores mean a worse outcome
change in dermatology life quality index (DLQI) | From enrollment to the end of treatment at 52 weeks
  range 0-30; higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Andreas Sygros Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsiogka A, Soulaidopoulos S, Gregoriou S, Rompoti N, Panagakis P, Papoutsaki M, Kostakis P, Kontochristopoulos G, Tsioufis K, Vlachopoulos C, Stratigos A, Rigopoulos D. Effects of IL17/23 Inhibitors on Markers of Subclinical Atherosclerosis in Patients with Psoriasis: An Observational Study. Dermatol Ther (Heidelb). 2025 Dec;15(12):3777-3792. doi: 10.1007/s13555-025-01549-1. Epub 2025 Oct 8. PMID 41060491

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT07169682/Prot_SAP_ICF_000.pdf